CLINICAL TRIAL: NCT07037420
Title: A Phase 2, Randomized, Double-blinded, Placebo-controlled, Dose Range-finding, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ALXN2420, a Growth Hormone Receptor Antagonist, Administered Subcutaneously in Combination With Somatostatin Analogs in Adult Participants With Acromegaly
Brief Title: ALXN2420 Versus Placebo in Combination With Somatostatin Analogs in Participants With Acromegaly
Acronym: ASTERIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7890C00001
Record Dates: First submitted 2025-05-27; First posted 2025-06-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acromegaly
Keywords: Acromegaly; ALXN2420; Somatostatin Analog; insulin-like growth factor 1; IGF-1; SSA therapy; GHRA; Growth Hormone Receptor Antagonist
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALXN2420 (Experimental): During the Primary Evaluation Period, participants will receive the first dose of ALXN2420 via SC injection on Day 1, followed by daily administration thereafter for a total of 15 weeks.
  Interventions: Drug: ALXN2420
- Placebo (Placebo Comparator): During the Primary Evaluation Period, participants will receive the first dose of placebo via SC injection on Day 1, followed by daily administration thereafter for a total of 15 weeks.
  Interventions: Drug: Placebo
- Open-label Extension Period (Experimental): During the Open-label Extension (OLE) Period, participants in the ALXN2420 treatment groups will continue receiving ALXN2420 treatment and participants in the placebo groups will crossover to receive ALXN2420 at Week 15. At the Week 15 Visit, the dose level and the dosing regimen of ALXN2420 will be determined for each participant based on the Week 13 IGF-1 level. The OLE Period assessments will be performed at Weeks 19, 26, 32, 39, 45, and 52.
  Interventions: Drug: ALXN2420

INTERVENTIONS:
Drug: ALXN2420 — ALXN2420 will be administered via subcutaneous (SC) injection
  Arms: ALXN2420; Open-label Extension Period
Drug: Placebo — Placebo will be administered via SC injection.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 15-week treatment with ALXN2420 versus placebo for decreasing insulin-like growth factor IGF-1 levels, when administered in combination with somatostatin analog (SSA) therapy to adult participants with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of acromegaly, that is, historically documented evidence of a GH-secreting pituitary adenoma based on MRI or pathology report
* Must be receiving maximum, or maximally tolerated dose per treating physician judgment, of long-acting SSAs (octreotide or lanreotide LAR) and meet both of the following:

  1. Received for ≥ 6 months prior to screening
  2. Receiving a once-monthly regimen (approximately every 4 weeks). Note: participants on stable regimens of other durations (for example, every 3 or 6 weeks) are not eligible
* Must be a partial responder to SSAs defined as > 20% relative IGF 1 reduction during the course of SSA therapy
* Serum IGF-1 levels > 1.3 to 5*ULN inclusive, as assessed at a central laboratory and adjusted for age and sex, based on average of 2 consecutive values obtained during the Screening Period and obtained ≥ 7 days apart

Exclusion Criteria:

* Had surgery for pituitary adenoma within the last 6 months before Day 1 or planning to receive surgery for pituitary adenoma during the study
* Pituitary adenoma that, per Investigator's judgment, is worsening as assessed by pituitary/sellar MRI or computed tomography scan obtained ≤ 6 months prior to screening
* Pituitary adenoma causing compression of the chiasm
* Clinical evidence of symptomatic hyperprolactinemia that would necessitate treatment with dopamine agonists
* Known hypothyroidism or hypocortisolism not adequately treated with a stable dose of thyroid or glucocorticoid hormone replacement therapy for ≥ 3 months prior to Screening
* Active, clinically significant cardiac disease as judged by the Investigator
* History of unstable angina, stroke, or acute myocardial infarction ≤ 3 months prior to screening
* Known uncontrolled type 2 diabetes (HbA1c > 10%)
* Active malignant disease ≤ 2 years prior to screening with exception of basal and squamous cell carcinoma of the skin
* Received any type of fractionated radiotherapy or a second surgical adenectomy for pituitary adenoma within the last 3 years (5 years for conventional radiation) before starting treatment and/or are planning to receive radiotherapy or a second surgical adenectomy during the study
* Received pegvisomant ≤ 8 weeks prior to screening
* Received dopamine agonists ≤ 4 weeks prior to screening
* Received pasireotide LAR ≤ 4 months prior to screening
* Clinically significant renal or hepatic disease at the time of screening, as judged by the Investigator
* eGFR (CKD-EPI formula) < 30 mL/minute/1.73 m^2 documented based on recent value (< 3 months prior to randomization)
* Clinically significant abnormal values for hematology, biochemistry, coagulation, or urinalysis, as judged by the Investigator, including, but not limited to, total bilirubin > 1.5*ULN (except if in free bilirubin linked to a known Gilbert Syndrome) or AST, ALT, or alkaline phosphatase > 2*ULN

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
Percentage Change From Baseline in Serum IGF-1 Level at Week 15 | Baseline, Week 15

SECONDARY OUTCOMES:
Number of Participants Who Achieve Serum IGF-1 Level ≤1.3 Upper Limit of Normal (ULN) at Week 15 | Week 15
Number of Participants Who Achieve of Serum IGF-1 Level ≤1.0 ULN at Week 15 | Week 15
Change from Basline in Symptoms as assessed by disease specific questionnaire, at Week 15 | Baseline, Week 15
Change From Baseline in Serum IGF-1 Level at Week 15 | Baseline, Week 15
Change From Baseline in 36-item Short Form Survey (SF-36) Summary Scores and Subscores at Week 15 | Baseline, Week 15
Change From Baseline in EuroQol 5-Dimension 5-Level (EQ-5D-5L) at Week 15 | Baseline, Week 15
Change From Baseline in Acromegaly Quality of Life (AcroQoL) at Week 15 | Baseline, Week 15
Change From Baseline in Global Impression of Severity at Week 15 as Assessed by Patient Global Impression of Severity (PGIS) Scale | Baseline, Week 15
Global Impression of Change at Week 15 as Assessed by Patient Global Impression of Change (PGIC) Scale | Week 15
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Adverse Events (AEs) Leading to Study Intervention Discontinuation or Interruption | Baseline (Day 1) through Week 15
Plasma Concentration of ALXN2420 | Baseline (Day 1) through Week 15
Number of Participants With Antidrug Antibodies (ADAs) | Baseline (Day 1) through Week 15

CONTACTS AND LOCATIONS:
Locations (41):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Torrance, California
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
- Argentina (2):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
- Brazil (4):
  - Research Site, Curitiba
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- China (4):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Kunming
  - Research Site, Shanghai
- Denmark (2):
  - Research Site, Copenhagen
  - Research Site, Odense
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Pécs
  - Research Site, Szeged
- Italy (7):
  - Research Site, Cona
  - Research Site, Genoa
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Netherlands (2):
  - Research Site, Leiden
  - Research Site, Rotterdam
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR